CLINICAL TRIAL: NCT05798260
Title: Intensive Care Unit (ICU) Biospecimen and Data Repository
Brief Title: T-Cell Mitochondrial Respiration Response to Ketone Monoester Supplement in Healthy Volunteers and COVID-19
Status: Withdrawn | Type: Observational
Why Stopped: Study Never Started
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00101196
Record Dates: First submitted 2023-03-28; First posted 2023-04-04 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: COVID-19 Acute Respiratory Distress Syndrome
Keywords: mitochondria; ketone monoester; seahorse; ketoneaid; SRC; FCCP; ECAR

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Volunteers: Healthy Volunteers
  Interventions: Diagnostic Test: Agilent Seahorse XF Cell Mito Stress Test
- COVID-19 positive admitted to the ICU and on the ventilator: COVID-19 positive admitted to the ICU and on the ventilator
  Interventions: Diagnostic Test: Agilent Seahorse XF Cell Mito Stress Test

INTERVENTIONS:
Diagnostic Test: Agilent Seahorse XF Cell Mito Stress Test — The Agilent Seahorse XF Cell Mito Stress Test measures key parameters of mitochondrial function by directly measuring the oxygen consumption rate (OCR) of cells on the Seahorse XFe and XF Extracellular Flux Analyzers. It is a plate-based live cell assay that allows to monitor spare respiratory capacity (SRC), basal respiration, ATP production-coupled respiration, maximal respiration, and non-mitochondrial respiration in real time before and after ketone monoester
  Other Names: Ketoneaid (Ketone monoester)

SUMMARY:
T-Cell Mitochondrial Respiration Response to Ketone monoester (Ketoneaid) in Healthy Volunteers and COVID-19

ELIGIBILITY:
Inclusion Criteria:

COVID-19 with ARDS and on the ventilator

Exclusion Criteria:

* Pregnant
* <18 years
* Steroid use

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients admitted at Duke Hospital Medical and Surgical ICU with COVID-19 manifested with ARDS and on the ventilator
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-06-30 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Spare Respiratory Capacity (SRC) | through study completion, an average of 2 months
  This measurement indicates the capability of the cell to respond to an energetic demand as well as how closely the cell is to respiring to its theoretical maximum. The cell's ability to respond to demand can be an indicator of cell fitness or flexibility
Basal Respiration | through study completion, an average of 2 months
  Oxygen consumption used to meet cellular ATP demand resulting from mitochondrial proton leak. Shows energetic demand of the cell under baseline conditions.
ATP production-coupled Respiration | upon admission
  The decrease in oxygen consumption rate upon injection of the ATP synthase inhibitor oligomycin represents the portion of basal respiration that was being used to drive ATP production. Shows ATP produced by the mitochondria that contributes to meeting the energetic needs of the cell.
Maximal Respiration | upon admission
  The maximal oxygen consumption rate attained by adding the uncoupler FCCP. FCCP mimics a physiological "energy demand" by stimulating the respiratory chain to operate at maximum capacity, which causes rapid oxidation of substrates (sugars, fats, and amino acids) to meet this metabolic challenge. Shows the maximum rate of respiration that the cell can achieve.
Non-Mitochondrial Respiration | through study completion, an average of 2 months
  Oxygen consumption that persists due to a subset of cellular enzymes that continue to consume oxygen after the addition of rotenone and antimycin A. This is important to get an accurate measure of mitochondrial respiration.

SECONDARY OUTCOMES:
Oxygen Consumption Rate (OCR) | through study completion, an average of 2 months
  The oxygen consumption rate (OCR) of cells is an important indicator of normal cellular function. It is used as a parameter to study mitochondrial function as well as a marker of factors triggering the switch from healthy oxidative phosphorylation to aerobic glycolysis
extracellular acidification rate (ECAR) | through study completion, an average of 2 months
  Measuring the extracellular acidification rate (ECAR) provides a method for detection of glycolytic flux in T-cells in response to ketone mono ester

CONTACTS AND LOCATIONS:
Overall Officials: Christina Barkauskas, MD, Principal Investigator — Research Director Duke Medical ICU
Locations (1):
- Christina Barkauskas, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No